CLINICAL TRIAL: NCT07172503
Title: Clinical Application of PET Imaging Targeting GPA33 in Malignant Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0907
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Gastric Cancer (GC); Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET imaging targeting GPA33 in malignant tumors (Experimental): Determine if targeting GPA33 PET is safe and effective method for imaging of malignant tumors.
  Interventions: Drug: 68Ga-NOTA-GPA33 nanobody

INTERVENTIONS:
Drug: 68Ga-NOTA-GPA33 nanobody — To perform integrated PET/MR or PET/CT visualization of patients with clinically suspected or confirmed colorectal cancer, gastric cancer, pancreatic cancer and other malignant tumors with high GPA33 expression and healthy volunteers, using specific positron imaging agents target GPA33(in the case of [68Ga]Ga-NOTA-GPA33 nanobody) , to achieve the following purposes: Patients with malignant tumors: for diagnosis and staging of diseases, comparing with the gold standard pathological diagnosis, evaluating diagnostic efficacy, clarifying the presence or absence of lesions, and determining the location and nature of lesions; comparing with [18F]FDG PET for accurate staging, evaluating the tumor load, and helping to determine the therapeutic plan. Healthy volunteers: Pharmacokinetic analysis will be performed to clarify the distribution and metabolism of the drug in the body and its safety.

SUMMARY:
This study is a diagnostic study. Patients and healthy volunteers with clinically suspected or confirmed colorectal cancer, gastric cancer, pancreatic cancer and other malignant tumors with high expression of GPA33 will be recruited for PET/MR or PET/CT imaging targeting a GPA33-specific probe (in the case of [68Ga]Ga-NOTA-GPA33 nanobody) , to observe the reaction of volunteers and patients after injection of drugs, to evaluate the pharmacokinetics in vivo and the efficacy of diagnosis and staging, and to perform PET imaging in patients with contraindications. General information on the subjects' vital signs, clinical data, blood routine, liver and kidney functions and other biochemical indicators and other imaging data were collected, and histopathology of biopsy or surgical specimens was used as the final diagnostic criterion.

DETAILED DESCRIPTION:
Malignant tumors are one of the major diseases leading to death worldwide, and their high incidence and mortality rates pose a serious threat to human health. According to the World Health Organization (WHO), there will be about 19.3 million new cancer cases and 10 million deaths globally in 2020, with a significant increase in the incidence of malignant tumors such as colorectal and gastric cancers in particular. Early diagnosis and load assessment of tumors are crucial for improving patient survival.Currently, there are limitations in the commonly used clinical diagnostic imaging tools. For example, traditional anatomical imaging techniques (e.g., ultrasound, CT, and MRI) have high resolution in displaying the anatomical structure of tumors, but it is difficult to accurately differentiate between benign and malignant lesions, and is not sufficiently sensitive to the performance of some tumors rich in fibrotic and necrotic tissues. Enhanced magnetic resonance imaging (ceMRI) has limited effectiveness in the detection of certain solid tumors, and is particularly deficient in the identification of microscopic lesions and some deep tumors. [18F]FDG PET/CT, a current widely used molecular imaging technique, enables functional imaging of tumors by reflecting the level of glucose metabolism. However, [18F]FDG is not a tumor-specific imaging agent, and non-malignant lesions such as inflammation, infection, and tuberculosis can also lead to an increase in local FDG uptake, producing false-positive results. In addition, [18F]FDG uptake is low in some tumors with low metabolic activity (e.g., poorly differentiated carcinomas and some brain tumors), leading to false-negative results and limiting its use in early tumor diagnosis and precision assessment. Therefore, the development of more specific and sensitive molecular imaging probes has significant clinical value. GPA33 is a member of the immunoglobulin superfamily, and as a novel transmembrane glycoprotein, it is significantly expressed in more than 95% of colorectal cancers, and mildly expressed in normal intestinal mucosa, as well as showing different degrees of expression in gastric and pancreatic cancers. Studies have shown that GPA33 has the functions of cell surface recognition and adhesion, as well as triggering intercellular signaling and immune response. These features make it has gradually become a potential marker for tumor diagnosis and treatment. In recent years, breakthroughs have been made in the research of targeted drugs against GPA33. However, how to screen patients suitable for targeted GPA33 therapy and dynamically evaluate the therapeutic effects remain clinical challenges. Therefore, the development of molecular imaging probes targeting GPA33 and the realization of non-invasive, real-time quantitative detection of GPA33 expression by PET imaging are expected to provide an imaging basis for targeted therapy. This can not only be used to screen patient groups with high GPA33 expression, thus accurately guiding the clinical application of targeted drugs, but also to assess drug efficacy in real time during the treatment process and promote the implementation of individualized treatment plans. In summary, the aim of this project is to explore the clinical application of PET imaging technology targeting GPA33 in malignant tumors, through PET imaging agents targeting GPA33 ([68Ga]Ga-NOTA-GPA33 nanobody as an example), with a view to be used for the diagnosis and staging of patients with malignant tumors, assessing the tumor load and the abundance of GPA33 expression, and assisting in the determination of the therapeutic regimen. Preliminary pharmacokinetic analysis was also performed in healthy volunteers to clarify the metabolic pattern and adverse effects of the drug in vivo.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all enrollment criteria to be eligible to participate in the study:

* 1: The subject or his/her legal representative is able to sign and date the informed consent form;
* 2: A commitment to comply with the research procedures and to cooperate in the implementation of the full research process;
* 3: Adult patients or healthy volunteers (aged 18 or above) of either sex;
* 4: Patients with clinically suspected or confirmed malignant tumors such as colorectal cancer, gastric cancer, pancreatic cancer (supporting evidence includes serum-related tumor markers, imaging data such as ultrasound, CT, MRI, etc., and histological pathology examination, etc.) and in good general condition;
* 5: Consistent with the results of specific laboratory tests;
* 6: Females of childbearing potential who have been using contraception for at least one month prior to screening and who are committed to using contraception for the entire study period and until a specified time after the end of the study；
* 7: Other set entry criteria.

Exclusion Criteria:

All subjects who meet any of the exclusion criteria baseline will be excluded from the study:

* 1: Those who are unable to complete a PET/MR or PET/CT examination (including inability to lie down, claustrophobia, radiophobia, etc.);
* 2: Having other comorbidities;
* 3: Patients with known hypersensitivity to GPA33 nanobody developers or synthetic excipients; fasting blood glucose level greater than 11.0 mmol/L prior to 18F-FDG injection；
* 4: Have a history of comorbid drug use;
* 5: Patients considered by the investigator to have poor compliance;
* 6: Patients during pregnancy or lactation;
* 7: Persons with other factors that make participation in this test inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual and standardized uptake values assessment of lesions and biodistribution | 1 year
  At least two experienced nuclear medicine physicians will conduct a visual analysis using consensus reading. The standardized uptake value (SUV) of tumor and organs will be measured after a semiquantitative analysis is conducted for each case. The SUV ranges from 0 to infinity, and a higher score means a higher uptake of targeting GPA33 nuclear probe by the tumor, which implies a greater threat of the tumor being malignant or higher stage.

SECONDARY OUTCOMES:
Radioactivity in the blood and urine samples | 1 year
  Blood samples were collected at 25 minutes, 55 minutes and 115 minutes after injection.
Pathological sections of tumour tissue | 1 year
  The excised tumour tissue was taken for immunohistochemistry to verify its GPA33 expression

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No